CLINICAL TRIAL: NCT03129542
Title: Oral Midodrine Hydrochloride in Early Sepsis: Randomized, Double Blind and Placebo-Controlled Feasibility Study
Brief Title: Midodrine Hydrochloride in Early Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Cleveland Clinic Abu Dhabi (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-002444
Record Dates: First submitted 2017-04-06; First posted 2017-04-26 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Sepsis; Blood Pressure
MeSH Terms: conditions — Sepsis | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: The Investigators propose a prospective, randomized, double blind, placebo-controlled pilot study on the efficacy and safety of midodrine in the treatment of sepsis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medical provider, nursing staff, study coordinator and patient will be blinded to randomization, only research pharmacist will be aware of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Midodrine Hydrochloride 10 milligrams (Active Comparator): Three doses of oral midodrine every 8 hours will be administered in addition to usual care for sepsis. Participants randomized to the intervention group will receive a total of 3 doses of midodrine 10 milligrams every 8 hours by mouth in the form of a tablet encapsulated in order to be identical to placebo. Participants will receive treatment for a total of 16 hours, beginning with the first dose.
  Interventions: Drug: Midodrine Hydrochloride 10 milligrams
- Placebo oral capsule (Placebo Comparator): For participants randomized to the placebo arm, an identical appearing capsule containing only Lactose Monohydrate powder will be administered every 8 hours for a total of 3 doses.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Midodrine Hydrochloride 10 milligrams — Three doses taken every 8 hours.
  Other Names: Midodrine
  Arms: Midodrine Hydrochloride 10 milligrams
Drug: Placebo capsule — Three doses taken every 8 hours.
  Other Names: Lactose Monohydrate powder
  Arms: Placebo oral capsule

SUMMARY:
The investigators would like to determine if early administration of oral Midodrine in participants diagnosed with sepsis will impact blood pressures and decrease the need for and/or doses of intravenous pressor agents.

DETAILED DESCRIPTION:
Three doses of either placebo or midodrine every 8 hours will be administered in addition to usual care for sepsis. The goal will be to administer the first dose approximately within 24 hours of diagnosis. The first dose will be administered only after the patient has been admitted to the ICU. Subjects will receive treatment for a total of 16 hours starting from the first dose. The medical provider, nursing staff and patient will be blinded to randomization, only research pharmacist will be aware of randomization. Blood pressure will be recorded at least on a 4 hourly basis for 24 hours from the time of administration of the first dose, and also just prior to administration of each dose. Subsequent doses will be held if systolic blood pressure, SBP, is greater than 130 mmHg. If a subject requires initiation of intravenous vasopressor agents following study enrollment, subsequent doses will be continued. There will be no further intervention after all 3 doses have been administered; however clinical outcomes and adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with sepsis based on the old Sepsis criteria and meeting all of the following criteria will be considered eligible to participate in the study.

* Age greater than or equal to 18 years
* Able to safely tolerate medication either by mouth or feeding tube (i.e. absence of nausea or vomiting)
* Able to give consent for participation or have representative available
* Two or more blood pressure readings taken at least 15 minutes apart with mean arterial pressures, MAPs 70 or less
* Treating consultant agrees to the study plan

Exclusion Criteria:

Patients meeting any one of the following criteria will be excluded from participation:

* Women of child bearing age with the potential to become pregnant who do not have a clinically documented negative pregnancy test
* Current cardiogenic shock or known systolic heart failure with left ventricular ejection fraction (LVEF) < 30%
* Current bowel ischemia
* Recent Myocardial infarction within the past 3 months
* Current use of Monoamine Oxidase Inhibitors (MAOIs)
* Recent Stroke within the past 3 months
* Midodrine as a home medication
* Known allergy to Midodrine
* High dose vasopressor use (norepinephrine >0.25 mcg/kg/min)
* Lactate more than 8 mmol/L
* Contraindications to use: History of pheochromocytoma or thyrotoxicosis or glaucoma or ischemic bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Duration of Vasopressor Use | 24 hours
  To study the duration of vasopressor use in the first 24 hours of sepsis

SECONDARY OUTCOMES:
Mean arterial blood pressure (MAP) | 24 hours after the first drug dose
  Routinely measured mean arterial blood pressure, invasive and noninvasive
Cumulative Fluid Balance | 24 hours after sepsis onset
  To study the cumulative fluid balance during the first 24 hours of sepsis
ICU and hospital length of stay, central venous access use and organ failure | The first 7 days of study enrollment or until discharge
  Daily Simplified Organ Failure Assessment, SOFA, scores
Incidence of potential side effects attributable to Midodrine | 48 hours after enrollment
  To study the potential side effects attributable to Midodrine use in diagnosis of Sepsis.
Cumulative Vasopressor Dose | 24 hours after the first drug dose
  To study the cumulative vasopressor dose requirements during the first 24 hours after study drug initiation

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Gajic, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials